CLINICAL TRIAL: NCT06486844
Title: Real World Outcomes of Patients Treated With Vericiguat in German Routine Care
Brief Title: An Observational Study Called ROVER to Learn More About How Well Vericiguat Works in People Who Were Newly Treated With Vericiguat in Routine Medical Care in Germany
Acronym: ROVER
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22829
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Chronic Heart Failure With Reduced Ejection Fraction
Keywords: HFrEF
MeSH Terms: interventions — vericiguat

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who received vericiguat prescription: Patients who were new users of vericiguat between September 2021 and September 2023 from the InGef database and the WIG2 database.
  Interventions: Drug: Vericiguat (Verquvo, BAY1021189)

INTERVENTIONS:
Drug: Vericiguat (Verquvo, BAY1021189) — Vericiguat was given following routine clinical practice.

SUMMARY:
This is an observational study in which data already collected from people treated with vericiguat are studied.

In observational studies, only observations are made without participants receiving any advice or any changes to healthcare.

Chronic heart failure with reduced ejection fraction (HFrEF) is a long-term condition that occurs when the heart is weak and cannot pump enough blood to the rest of the body with each heartbeat. This leads to a reduced supply of oxygen which the body requires to function properly. The common symptoms include breathlessness, weakness, fatigue, and swelling in the ankles and legs. If left untreated, heart failure can lead to other serious health problems, including damage to other organs, which may result in hospital stays and even death.

Vericiguat works by increasing the activity of an enzyme called soluble guanylate cyclase (sGC), which relaxes the blood vessels and allows more blood to flow through. As a result, the heart is able to pump better.

Vericiguat is available in Germany for the treatment of HFrEF based on the results of a study called VICTORIA. The VICTORIA study showed that vericiguat helps in lowering the chances of death or hospitalization due to heart failure. However, there is limited information available about the use of vericiguat for the treatment of HFrEF under real-world conditions in routine medical care.

The main purpose of this study is to collect information about how well vericiguat works in people with HFrEF who were newly treated with vericiguat. In addition, researchers will collect information about participants' basic characteristics, including their age, gender, other health conditions they might have, and the medicines they might be taking.

The data will come from 2 German health databases including people who newly started vericiguat treatment between September 2021 and September 2023.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an initial prescription of Vericiguat (index date) according to ATC Code C01DX22.
* At least 18 years or older on the initial prescription of Vericiguat.

Exclusion Criteria:

* No exclusion criteria for any population will be applied.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with their first vericiguat prescription since market authorization in September 2021 who are aged 18 years or older will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2024-07-05 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
All-cause mortality rates after initiation of vericiguat | Between September 2021 and September 2023
  Number of patients who died between the "Vericiguat index date" and "cohort exit" according to their death date.
All-cause related hospitalization rates after initiation of vericiguat | Between September 2021 and September 2023
  Sum of all fully hospitalized cases of all patients between the "Vericiguat index date" and "cohort exit".
Heart failure related hospitalization rates after initiation of vericiguat | Between September 2021 and September 2023
  Sum of all fully hospitalized cases with a main or secondary inpatient diagnosis according to ICD-10 GM Code I50.x or I11.0 between the "Vericiguat index date" and "cohort exit".

SECONDARY OUTCOMES:
Adherence of vericiguat drug use | Between September 2021 and September 2023
  Adherence will be assessed using the Medical Possession Ratio (MPR=days of supply/treatment duration).
Titration pattern of vericiguat drug use | Between September 2021 and September 2023
  Titration patterns will be assessed by investigating indicators such as the starting dose, the maximum dose reached as well as the time until up-titration.
Patient persistence of vericiguat drug use | Between September 2021 and September 2023
  Persistence will be calculated via the time until discontinuation of vericiguat.
Socio-demographic characteristics of patients initiating vericiguat at baseline | Between September 2021 and September 2023
  Sex and age groups.
Clinical characteristics of patients initiating vericiguat at baseline | Between September 2021 and September 2023
  Pre-defined comorbidities, pre-defined comedications, all-cause hospitalization, worsening hart failure event, etc.
Medication of interest in the 3 months before and after initiation of vericiguat | Between September 2021 and September 2023

CONTACTS AND LOCATIONS:
Locations (1):
- Bayer, Wuppertal, Germany

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.